CLINICAL TRIAL: NCT06550583
Title: A Clinical Audit on Screening Program for Early Cervical Cancer Detection.
Brief Title: Screening for Early Cervical Cancer Detection
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Abdelraof Soliman, Principal investigator, Assiut University
Other Study IDs: screening for cervical cancer
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cervical Cancer; Cervix Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Pap smear test results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pap smear /Test — Patients will be placed in the lithotomy position, and a sterile bivalve speculum will be inserted into the vagina.
  • A sample will be taken from the ectocervix by rotating a wooden Ayre spatula 360°. The sample will be quickly smeared onto a labeled glass slide and fixed with 95% ethyl alcohol in a jar to be sent to the Department of Pathology for cytopathological examination

SUMMARY:
This study is to audit results and adherence to Cervical Screening program before and after the implementing awareness of the WHO guidelines of screening among the multidisciplinary healthcare workers and patients.

DETAILED DESCRIPTION:
Cervical cancer screening is the asymptomatic detection of pre-cancer and cancer in women at risk, with at least one screening suggested for women aged 30-49 years. According to the World Health Survey (2015), 19% of eligible women in developing countries and 63% of those in developed nations had their cervical cancer screening done using a Pap smear or visual inspection with acetic acid (VIA).

According to latest estimates by World Health Organization (WHO), in Egypt, 866 women are diagnosed with cervical cancer every year and 373 die from the disease. Cervical cancer is the 13th most common cancer in women in Egypt and the 10th most common cancer in women aged between 15 to 44 years . Statistics from Egyptian studies provide pre invasive cervical lesion incidence levels of 0.3 % to 0.5 % .

The human papillomavirus (HPV) is one of the most significant risk factors for cervical cancer. HPV can be transmitted through sexual contact, including vaginal or oral sex with an infected person. HPV has more than 100 strains, of which HPV16 and HPV18 account for about 70% of invasive cervical cancers

ELIGIBILITY:
Inclusion Criteria:

* Women 20-60 years.

  * Sexually active.
  * Fulfilling Cervical Check's eligibility criteria for screening at the time of the audit https://www.cervicalcheck.ie/_fileupload/File/Eligibility%20Framework.pdf

Exclusion Criteria:

Patient who had underwent to total hysterectomy.

* Pregnant or postpartum or post abortive patients
* Patient having any history of treatment for cervical dysplasia.
* Immunocompromised patients.

Ages: 20 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — sexually active women in reproductive age .
Study Population: Female patients who will attend gynecology clinics at Women & Children Hospital in reproductive age in (Assuit) Egypt
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Screening clinic in Women & Children Hospital | Baseline
  All women undergo Pap smear test according to inclusion criteria and will be adherence to screening program protocol

SECONDARY OUTCOMES:
Via test | baseline
  Via test will be done to all patients come to screening clinic and Adherence to screening program protocol

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Soliman, physician, Study Chair — Assiut University; Hisham A Alsayed Abotaleb, professor, Study Director — Assiut University; Hazem S Eldeen Mohammed, professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Amado G, Weldegebreal F, Birhanu S, Dessie Y. Cervical cancer screening practices and its associated factors among females of reproductive age in Durame town, Southern Ethiopia. PLoS One. 2022 Dec 30;17(12):e0279870. doi: 10.1371/journal.pone.0279870. eCollection 2022. PMID 36584208
- [Background] Attallah O. Cervical cancer diagnosis based on multi-domain features using deep learning enhanced by handcrafted descriptors. Applied Sciences. 2023;13(3):1916.
- [Background] Burmeister CA, Khan SF, Schafer G, Mbatani N, Adams T, Moodley J, Prince S. Cervical cancer therapies: Current challenges and future perspectives. Tumour Virus Res. 2022 Jun;13:200238. doi: 10.1016/j.tvr.2022.200238. Epub 2022 Apr 20. PMID 35460940
- [Background] Hakimi S, Lami F, Allahqoli L, Alkatout I. Barriers to the HPV vaccination program in the Eastern Mediterranean region: a narrative review. J Turk Ger Gynecol Assoc. 2023 Mar 15;24(1):48-56. doi: 10.4274/jtgga.galenos.2022.2022-6-6. Epub 2022 Dec 30. PMID 36583290
- [Background] Haran M, Kelly JR, Kennedy L, Hennigan K, Farid H, Herteu C, Kreisel A, Salehin S, O' Sullivan M, Keating S, Ivers JH, Scully M. An audit of the cervical screening programme in the National Drug Treatment Centre (NDTC). Ir J Med Sci. 2021 Nov;190(4):1379-1386. doi: 10.1007/s11845-020-02459-1. Epub 2021 Jan 15. PMID 33449334
- [Background] Mohammed MS, Sand AS, Hassuna NA. Prevalence of HPV 16 and HPV 18 in cervical cancer in Minia Governorate. Egyptian Journal of Medical Microbiology. 2020;29(4):57-63.
- [Background] Momenimovahed Z, Mazidimoradi A, Maroofi P, Allahqoli L, Salehiniya H, Alkatout I. Global, regional and national burden, incidence, and mortality of cervical cancer. Cancer Rep (Hoboken). 2023 Mar;6(3):e1756. doi: 10.1002/cnr2.1756. Epub 2022 Dec 21. PMID 36545760
- [Background] Nayar R, Wilbur DC. The Bethesda System for Reporting Cervical Cytology: A Historical Perspective. Acta Cytol. 2017;61(4-5):359-372. doi: 10.1159/000477556. Epub 2017 Jul 11. PMID 28693017
- [Background] Nilima N, Mani K, Kaushik S, Rai SN. Cervical Cancer Screening and Associated Barriers among Women in India: A Generalized Structural Equation Modeling Approach. Cancers (Basel). 2022 Jun 23;14(13):3076. doi: 10.3390/cancers14133076. PMID 35804848
- [Background] Romli R, Abd Rahman R, Chew KT, Mohd Hashim S, Mohamad EMW, Mohammed Nawi A. Empirical investigation of e-health intervention in cervical cancer screening: A systematic literature review. PLoS One. 2022 Aug 19;17(8):e0273375. doi: 10.1371/journal.pone.0273375. eCollection 2022. PMID 35984812
- [Background] Wang J, Elfstrom KM, Andrae B, Nordqvist Kleppe S, Ploner A, Lei J, Dillner J, Sundstrom K, Sparen P. Cervical cancer case-control audit: Results from routine evaluation of a nationwide cervical screening program. Int J Cancer. 2020 Mar 1;146(5):1230-1240. doi: 10.1002/ijc.32416. Epub 2019 Jun 3. PMID 31107987
- [Background] Zhu J, Ge Z, Xia J, Liu Q, Ran Q, Yang Y. Status quo and problem analysis of cervical cancer screening program in China: Based on RE-AIM framework. Front Public Health. 2022 Oct 14;10:987787. doi: 10.3389/fpubh.2022.987787. eCollection 2022. PMID 36311598